CLINICAL TRIAL: NCT01045187
Title: Feasibility Study Using the Xoft Axxent Electronic Brachytherapy System for the Treatment of Endometrial Cancer
Brief Title: Feasibility Study Using the Xoft System for the Treatment of Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xoft, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR-0209
Record Dates: First submitted 2009-11-19; First posted 2010-01-08 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; Uterine cancer; electronic brachytherapy; Xoft
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — Brachytherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endometrial cancer (Other): Patients are treated with electronic brachytherapy for an FDA cleared indication.
  Interventions: Radiation: brachytherapy; Radiation: Xoft Axxent Electronic Brachytherapy System

INTERVENTIONS:
Radiation: brachytherapy — Electronic brachytherapy dose 21 Gy or 22 Gy in 3-4 fractions prescribed to 5mm depth, or electronic brachytherapy 16-18 Gy if EBRT is administered.
  Other Names: Electronic; Radiation; Vaginal cuff
Radiation: Xoft Axxent Electronic Brachytherapy System — 21-22 Gy in 3-4 fractions to 5mm or 16-18 Gy in 3 fractions prescribed to the surface.
  Other Names: Radiation; therapy; electronic

SUMMARY:
Multicenter, non-randomized, feasibility study to evaluate the treatment and assess acute safety of the FDA Cleared Axxent Electronic Brachytherapy System and vaginal applicator for intracavitary vaginal cuff treatment according to the physician's current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Most types of endometrial (uterine) cancer Stage I and Stage II (see exclusion criteria below)
* Post hysterectomy

Exclusion Criteria:

* Endometrial (uterine) cancer Stage IA Grade 1
* Scleroderma
* Collagen vascular disease
* Active Lupus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dickler, MD, Principal Investigator — Little Company of Mary
Locations (6):
- United States (6):
  - Cancer Treatment Services Arizona, Casa Grande, Arizona
  - Southwest Oncology Center, Phoenix, Arizona
  - Beverly Oncology & Imaging Medical Center, Inc, Montebello, California
  - Swedish Covenant Hospital, Chicago, Illinois
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Dickler A, Puthawala MY, Thropay JP, Bhatnagar A, Schreiber G. Prospective multi-center trial utilizing electronic brachytherapy for the treatment of endometrial cancer. Radiat Oncol. 2010 Jul 20;5:67. doi: 10.1186/1748-717X-5-67. PMID 20646289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from September 2008 through October 2009. The centers were at Hospitals and free-standing radiation oncology clinics.
Pre-assignment Details: Patients who were candidates for vaginal brachytherapy post TAH-BSO with or without EBRT were enrolled. Patient participation was voluntary for this data collection study.
Period: Overall Study
Arm/Group | Endometrial Cancer
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endometrial Cancer
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Assess Number of Patients Who Were Able to Complete Treatment Delivery Using the Axxent Electronic Brachytherapy System
Time Frame: through completion of radiation therapy
Measure: Number; unit: Participants
Arm/Group | Endometrial Cancer
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Assess Acute Safety Outcomes in Patients During and After Vaginal Cuff Brachytherapy Treatment With the Axxent Electronic Brachytherapy System as Incorporated in to the Physician's Current Standard of Practice
Time Frame: through 3 month post treatment
Reporting Status: Not Posted

3. Secondary Outcome: Assess Occurence Rate of Toxicities
Time Frame: through 3 month follow up post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Procedure through 3 month follow-up to report acute toxicities.
Arm/Group | Endometrial Cancer
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cancer (N=15)
Dysuria (Renal and urinary disorders) | 2 (2) — Dysuria Grade 1 at 1 month ongoing at 3 months. Dysuria grade 2 at 1 month resolved at 3 months.
Pain (Reproductive system and breast disorders) | 1 (1) — Occurrence rate= 1 patient at 1 visit: Vaginal pain grade 2 t 1 month resolved at 6 weeks.
Mucosal Atrophy (Reproductive system and breast disorders) | 1 (1) — Reported x 1: Mucosal atrophy grade 1 reported at 3 month visit and noted to be resolved at 3 month visit.
Rectal bleeding (Gastrointestinal disorders) | 1 (1) — Grade one reported at 3 month visit and noted to be resolved at that time.
Vaginal drying (Reproductive system and breast disorders) | 1 (1) — Vaginal Drying grade one reported x 1 at 3 months and oted to be resolved at 3 months.

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No